CLINICAL TRIAL: NCT03837457
Title: PRISM: An Open-label, Multi-Center Extension Study to Investigate the Efficacy and Safety of Cobomarsen (MRG-106) Following Systemic Treatment in Subjects With Cutaneous T-Cell Lymphoma (CTCL), Mycosis Fungoides (MF) Subtype, Who Have Completed the SOLAR Study
Brief Title: PRISM: Efficacy and Safety of Cobomarsen (MRG-106) in Subjects With Mycosis Fungoides Who Have Completed the SOLAR Study
Acronym: PRISM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study no longer needed because eligible subjects may receive treatment with cobomarsen in a crossover arm of the SOLAR clinical trial (NCT03713320)
Sponsor: miRagen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG106-11-203; 2018-003748-22 (EudraCT Number)
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Cutaneous T-Cell Lymphoma/Mycosis Fungoides
Keywords: PRISM; Cutaneous T-cell Lymphoma; CTCL; Mycosis Fungoides; Lymphoma; Lymphoma, T-cell; Lymphoma, T-cell, cutaneous; Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Neoplasms; MicroRNAs
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous; Lymphoma; Lymphoma, T-Cell; Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Neoplasms | interventions — cobomarsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cobomarsen (Experimental)
  Interventions: Drug: Cobomarsen

INTERVENTIONS:
Drug: Cobomarsen — At least weekly intravenous infusions of cobomarsen (282 mg) throughout study treatment period
  Other Names: MRG-106

SUMMARY:
The main objective of this clinical trial is to study the efficacy and safety of cobomarsen (also known as MRG-106) for the treatment of cutaneous T-cell lymphoma (CTCL), mycosis fungoides (MF) subtype in subjects who have confirmed disease progression following treatment with vorinostat in the SOLAR clinical study (MRG106-11-201). Cobomarsen is designed to inhibit the activity of a molecule called miR-155 that may be important to the growth and survival of MF cancer cells.

The effects of treatment will be measured based on changes in skin lesion severity, disease-associated symptoms, and quality of life, as well as the length of time that the subject's disease remains stable or improved, without evidence of disease progression. The safety and tolerability of cobomarsen will be assessed based on the frequency and severity of observed side effects.

DETAILED DESCRIPTION:
Study Design:

Up to 60 subjects are expected to be enrolled after discontinuation from the SOLAR clinical study (MRG106-11-201). Cobomarsen will be administered in the clinic by 2-hr intravenous infusion on Days 1, 3, 5 and 8, and weekly thereafter. Treatment will continue until the subject becomes intolerant, develops clinically significant side effects, progresses, or the trial is terminated.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have participated in the comparator arm of the SOLAR clinical trial and completed the study (confirmed disease progression).

Key Exclusion Criteria:

* Sézary syndrome or mycosis fungoides with B2 involvement, defined as documented history of B2 and/or B2 staging at screening.
* Evidence of large cell transformation.
* Visceral involvement related to MF at screening.
* Unresolved toxicities from prior vorinostat treatment, defined as having not resolved to CTCAE v5.0 grade 0 or 1.
* Any CTCL systemic therapy after completion of the SOLAR study and prior to Day 1 for PRISM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving an objective response of at least 4 months duration (ORR4) | Up to approximately 36 months (estimated study duration)
  Based on composite global response criteria including radiological imaging, flow cytometry, and the modified Severity Weighted Assessment Tool (mSWAT).

SECONDARY OUTCOMES:
Progression-free survival | Up to approximately 36 months (estimated study duration)
  Time from date of first dose of cobomarsen until the date of earliest documented progression or death from any cause.
Pruritis Numerical Rating Scale | Daily for up to 6 months, then weekly up to approximately 36 months (estimated study duration)
  Measures the patient's degree of itch related to mycosis fungoides based on an 11-point scale (from 0-10), with 0 being no itch and 10 being worst imaginable itch.
Skindex-29 Dermatological Survey | Monthly, up to approximately 36 months (estimated study duration)
  Measures the effects of skin disease on quality of life based on a 30-item questionnaire. The patient's responses are transformed to a linear scale from 0 to 100 and averaged to determine a subscore in three domains (Symptoms, Emotions and Functioning), as well as a total score. Lower scores indicate a lesser degree of skin disease interference with quality of life.
Pain Numerical Rating Scale | Daily, for up to 6 months, then weekly up to approximately 36 months (estimated study duration)
  Measures the patient's intensity of pain related to mycosis fungoides based on an 11-point scale (from 0-10), with 0 being no pain and 10 being worst imaginable pain.
Difference in drug tolerability by Patient Impression of Treatment Side Effects | Weekly, up to approximately 36 months (estimated study duration)
Duration of composite global response for responding subjects | Up to approximately 36 months (estimated study duration)
Complete response rate | Up to approximately 36 months (estimated study duration)
  Based on composite global response criteria including radiological imaging, flow cytometry, and mSWAT.
Skin disease severity based on modified Severity-weighted Assessment Tool (mSWAT) | Monthly, up to approximately 36 months (estimated study duration)
  Measures skin disease severity based on the percentage of skin within each body region with patches, plaques, or tumors. Total scores are calculated by adding the total percent for each category of lesion (patch, plaque, or tumor) and multiplying by a weighting factor. Weighted subtotals are added together to obtain the total score. Lower scores indicate a lower degree of skin disease severity.
Time to progression | Up to approximately 36 months (estimated study duration)
  Time from date of first dose of cobomarsen until the earliest date of confirmed progression.
Overall survival | Up to approximately 36 months (estimated study duration)
  Time from date of first dose of cobomarsen until the date of death from any cause.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to approximately 36 months (estimated study duration)
Plasma concentration of cobomarsen | Day 1, Day 29 and monthly or every other month thereafter until End of Treatment visit, up to approximately 36 months (estimated study duration)
  Sparse pharmacokinetic samples will be collected to monitor for accumulation of cobomarsen.

OTHER OUTCOMES:
Number of participants with anti-drug antibody generation | Up to approximately 36 months (estimated study duration)

CONTACTS AND LOCATIONS:
Overall Officials: Diana M. Escolar, MD, FAAN, Study Director — miRagen Therapeutics, Inc.
Locations (9):
- United States (5):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - The Ohio State University and Wexner Medical Center, Columbus, Ohio
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington
- University Hospital Leuven, Leuven, Belgium
- France (3):
  - Hopital Saint Andre, CHU de Bordeaux, Bordeaux
  - Hopital Saint-Louis, Paris
  - Hopital Charles Nicolle, CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No